CLINICAL TRIAL: NCT02401581
Title: Study ¨PRECOCE Feasibility Study of Photovaporisation of Prostate With a Limitated Length of Catheterization of 3 Hours
Brief Title: Feasibility Study of Photovaporisation of Prostate With a Limitated Length of Catheterization of 3 Hours
Acronym: PRECOCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-PP-07
Record Dates: First submitted 2014-12-01; First posted 2015-03-30 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Benign Prostatic Hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rate of early removal of the catheter (Experimental): In our study, we propose to evaluate the failure rate of an early removal of the catheter 3 hours post-operative after a PVP procedure with GL 180 W/XPS in selected patients on general anesthesia or spinal anesthesia for limiting autonomic effects on the bladder and ensure fastest possible recovery of voiding .
  Interventions: Other: Catheter

INTERVENTIONS:
Other: Catheter — The effectiveness of this model of management is defined by absence of a need for re-catheterization in the post -operative period of 24 hours, indications for resondage being cases of acute urinary retention (AUR ) or macroscopic hematuria necessitating a washes with drainage . Patients are followed for a period of 3 months with a post-operative visit at 30 days and a last follow-up visit at 90 days during which the effectiveness is evaluated by conventional means of clinical indicators ( flowmetry , postvoid residue, volumetry of the prostate , IPSS scores , QoL , EVA, IIEF ... ).

SUMMARY:
Benign hypertrophy of the prostate (BPH) is the most frequent pathology in the urinary tract of middle-aged men. In recent years, to enable BPH treatment with larger volumes and to reduce the risk of hemorrhage known to be associated to the transurethral resection of prostate treatment, transurethral photovaporisation of the prostate (PVP ) with the GreenLight (GL) XPS 180 W was developed. Therefore, the question arises to maximally reduce the length of catheterization to facilitate outpatient surgical management of prostate adenoma.

In the investigators study, the investigators propose to evaluate the failure rate of an early removal of the catheter 3 hours post-operative after a PVP procedure with GL 180 W/XPS in selected patients on general anesthesia or spinal anesthesia. To this end, the investigators realize a national multicenter prospective study including 300 patients. The effectiveness of this model of management is defined by absence of a need for re-catheterization in the post -operative period of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. patients with lower urinary tract symptoms (LUTS )
2. IPSS≥ 15 despite medical treatment > 1 month if monotherapy or > 3 months if bitherapie OR acute urinary retention ( RAU ) non-medical after the 1st failure to remove the catheter OR acute prostatitis OR macroscopic haematuria of prostatic origin
3. prostate volume > 30 cc by transrectal ultrasonography ;
4. IPSS Qol ≥ 3 has at inclusion ;
5. PSA ≤ 4 ng / ml ;
6. if PSA between 4 and 10 then PSA L/T ≥25 % or negative PBP <6 months .
7. Accommodation <50 km;
8. company available for the return at home and monitoring first post- operative night .
9. patient sign the informed consent
10. patient covered by social security or other health insurance

Exclusion criteria

1. post- voiding residue > 250 cc by suprapubic ultrasound not older than < 45 days
2. prostate volume > 100 cc by transrectal ultrasound not older than 45 days
3. urological antecedents : o urethral stenosis or cervical disease

   * UTI in progress
   * SAD patient or self-catheterization
   * obstructive hydronephrosis + / - renal failure
   * vesical calculi
   * cancer of the prostate treated or untreated
   * bladder tumor associated
   * Interstitial cystitis ( symptom or biopsy)
4. antecedent of the prostate surgery
5. neurologic bladder ( parkinsonian syndrome , multiple sclerosis , lupus, neuropathy, Diabetic, cauda equina syndrome )
6. criteria related concomitant medications that can not be stopped at least < 48 hours before PVP with GL XPS 180 W
7. contra indication for outpatient care for medical reason
8. contra indication of a product analgesic according to protocol
9. patient inability to understand and sign the informed consent as well as completing the questionnaires
10. ASA Score > 3 .

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
failure rate of a limited catheterization duration of 3 hours post- operative | at three hours post surgery
  • The failure rate of a limited catheterization duration of 3 hours post- operative is defined by a need of recatheterizatrion within 24 hours post- GL with PVP XPS 180W . The catheterization remains indicated in case of macroscopic hematuria RAU or if no natural urination is possible

SECONDARY OUTCOMES:
Total dose of energy | during 24 hours hospitalisation
  The total dose of energy delivered to the tissue induring the intervention will be expressed and collected by means of the instrumentation of the GL-XPS console.
The duration of recatherization | during 24 hours hospitalisation
  The duration of recatherization is regarded as the total cumulative duration of catheterization regardless of the number of attempts for removale when it is a failure. The average duration of resondage counts only recatheterizations occurring in the first week which may be considered as due to PVP with GL XPS 180W followed by a shortened catheterization of 3 hours post- operatively . The duration of recatherization is defined from the time when it was done in thefirst week post- operative until urinary recovery

CONTACTS AND LOCATIONS:
Overall Officials: DURAND Matthieu, Ph, Principal Investigator — Service d'Urologie, CHU de Nice
Locations (12):
- France (12):
  - CH Grasse - urologie, Grasse, Alpes-maritimes
  - CHU de Nice - Urologie, Nice, Alpes-Maritimes
  - CH privé St Brieuc, Saint-Brieuc, Cote D'armor
  - APHM - Urologie - Hôpital Conception, Marseille, PACA
  - CHRU Tours, Tours, Vendée
  - CHU Brest Urologie, Brest
  - CHU Grenoble, Grenoble
  - CHU Limoges -Urologie - Hôpital Dupuytren, Limoges
  - Polyclinique les Bleuets, Reims
  - CHU Rennes, Rennes
  - AP-HP - Urologie Hôpital Tenon, Paris, Île-de-France Region
  - Institut Mutualiste Monsouris urologie, Paris, Île-de-France Region